CLINICAL TRIAL: NCT04761757
Title: Antidepressant Decision Aid for Major Depressive Disorder Patients
Acronym: ADAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Collaborators: Ministry of Education, Malaysia (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ADAM
Record Dates: First submitted 2021-01-24; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Depression; Depressive Symptoms; Depressive Disorder, Major; Mood Disorders
Keywords: Shared decision making; Patient decision aid
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Mood Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Active Comparator)
  Interventions: Other: Booklet of Scripts of Doctors
- Intervention Arm (Active Comparator)
  Interventions: Other: Booklet of Scripts for Doctors and the Antidepressant Decision Aid for Major depressive disorder patients (ADAM)

INTERVENTIONS:
Other: Booklet of Scripts of Doctors — The "Booklet of Scripts for Doctors" was used in the control arm. This tool was developed and tested to encourage shared decision-making in prescribing antidepressants within the Malaysian context.
  Arms: Control Arm
Other: Booklet of Scripts for Doctors and the Antidepressant Decision Aid for Major depressive disorder patients (ADAM) — The "Booklet of Scripts for Doctors" along with the "Antidepressant Decision Aid for Major depressive disorder patients, ADAM", was used in the intervention arm. The decision aid was developed as per the International Patient Decision Aid Standards (IPDAS) criteria to enhance patient understanding of risks and benefits of different antidepressants available within the Malaysian context.
  Arms: Intervention Arm

SUMMARY:
The purpose of this study is to determine whether Antidepressant Decision Aid for Major Depressive Disorder is feasible and effective in involving patients in the decision-making process when initiating pharmacotherapy.

DETAILED DESCRIPTION:
To examine the ability of the patient decision aid to enhance shared decision making and preparedness to make decisions pertaining to antidepressant therapy. The research team has systematically developed an Antidepressant Decision Aid for Major depressive disorder patients (ADAM) according to the International Patient Decision Aids Standards (IPDAS) and the Ottawa Decision Support Framework. This is a posttest-only study with nonequivalent groups to evaluate the effect of the antidepressant decision aid on patient and physician perception of shared decision making as well as patient preparedness for making pharmacotherapeutic decisions compared usual care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Major Depressive Disorder (MDD)
* No psychotic symptoms
* Based on psychiatrist's clinical judgement currently in need for antidepressant treatment.
* Functional English literacy and language skills (to use the decision aid and fill out the questionnaires)
* Provides consent

Exclusion Criteria:

* Psychosis
* Communication barriers (visual impairment, language barrier)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 752 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Shared Decision Making_Patient Perspective | Immediately after the clinical encounter
  The patient version of the Shared Decision Making scale (SDM-Q-9) measures the extent to which patients are involved in the decision-making process from the patient's perspective. It consists of nine items rated on a six-point Likert-type scale from"completely disagree=" to"completely agree=". Adding the score of all the items leads to a raw total between 0 and 45. Multiplying the raw score by 20/9 provides a transformed score ranging from 0 to 100, higher scores indicate a greater extent of SDM.
Shared Decision Making_Physician Perspective | Immediately after the clinical encounter
  The physician version of Shared Decision Making scale (SDM-Q-Doc) measures the extent to which patients are involved in the decision-making process from the physician's perspective. It consists of nine items rated on a six-point Likert-type scale from"completely disagree=" to"completely agree=". Adding the score of all the items leads to a raw total between 0 and 45. Multiplying the raw score by 20/9 provided a transformed score ranging from 0 to 100, higher scores indicate a greater extent of SDM.
Preparation for Decision Making_Patient Perspective | Immediately after the clinical encounter
  The patient version of the Preparation for Decision-Making Scale (PDMS) assesses the patient's perception of how the PDA helped them recognize that a decision needs to be made, preparing them to communicate with their practitioner and promote patient involvement in the decision-making process. Higher scores indicate a higher perceived level of preparation for decision making.
Preparation for Decision Making_Physician Perspective | Immediately after the clinical encounter
  The physician version of the Preparation for Decision-Making Scale (PDMS) assesses the physician's perception of how the PDA helped patients recognize that a decision needs to be made, preparing them to communicate with their practitioner and promote patient involvement in the decision-making process. Higher scores indicate a higher perceived level of preparation for decision making.

CONTACTS AND LOCATIONS:
Overall Officials: Aya Ahmed Abousheishaa, Principal Investigator — University of Malaya; Ng Chong Guan, Principal Investigator — University of Malaya
Locations (17):
- Malaysia (17):
  - Columbia Asia Hospital, Iskandar Puteri, Johor
  - Hospital Permai, Johor Bahru, Johor
  - Sultanah Aminah Hospital, Johor Bahru, Johor
  - KPJ Ampang Puteri Specialist Hospital, Ampang, Kuala Lumpur
  - Dr Seed Specialist Clinic, Kepong, Kuala Lumpur
  - Hospital Pengajar Universiti Putra Malaysia, Serdang, Kuala Lumpur
  - Hospital Sultan Haji Ahmad Shah, Temerluh, Pahang
  - Hospital Raja Permaisuri Bainun, Ipoh, Perak
  - Hospital Pulau Pinang, George Town, Pulau Pinang
  - Hospital Umum Sarawak, Kuching, Sarawak
  - A. H. Lee Specialist Clinic, Petaling Jaya, Selangor
  - Hospital Sultanah Nur Zahirah, Kuala Terengganu, Terengganu
  - Hospital Pusrawi, Kuala Lumpur
  - Klinik Pakar Dr Yeoh & Dr Hazli Mental Health Specialist, Kuala Lumpur
  - Pusat Perubatan Universiti Kebangsaan Malaysia, Kuala Lumpur
  - University of Malaya Medical Centre, Kuala Lumpur
  - Hospital Putrajaya, Putrajaya

IPD SHARING:
Plan to Share IPD: No